CLINICAL TRIAL: NCT04933916
Title: Efficacy and Safety of Combination EMB-001 as a Potential Smoking Cessation Treatment
Brief Title: Study of EMB-001 as a Potential Smoking Cessation Treatment
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Business decision
Sponsor: Embera NeuroTherapeutics, Inc. (Industry)
Collaborators: Foundation for a Smoke Free World INC (Other); Rose Research Center, LLC (Industry); Segal Trials (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ERL-T002
Record Dates: First submitted 2021-06-14; First posted 2021-06-22 (Actual); Last update posted 2023-08-09 (Actual); Status verified 2023-08

CONDITIONS: Tobacco Use Disorder
Keywords: smoking; tobacco use; smoking cessation
MeSH Terms: conditions — Tobacco Use Disorder; Smoking; Tobacco Use; Smoking Cessation

STUDY DESIGN:
Intervention Model Description: Open-label
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- EMB-001 Active (Experimental): 720 mg metyrapone/24 mg oxazepam mg BID, for a total daily dose of 1440 mg metyrapone and 48 mg oxazepam
  Interventions: Drug: EMB-001

INTERVENTIONS:
Drug: EMB-001 — Combination product metyrapone and oxazepam

SUMMARY:
EMB-001 is a combination of 2 drugs: the cortisol synthesis inhibitor, metyrapone (Metopirone®), and the benzodiazepine receptor agonist, oxazepam (original trade name Serax®; now marketed as oxazepam (generic) only).

This is an open-label study in up to 50 adult subjects to help smokers abstain from smoking during a 12-week trial period.

DETAILED DESCRIPTION:
This an exploratory, single-group, open-label study of up to 50 subjects to evaluate the effects on smoking cessation and the safety and tolerability of EBM-001 in smokers.

After obtaining informed consent, adult smokers will be enrolled into the study. There will be an observational period of at least five days to obtain baseline data on use of combustible cigarettes.

Subjects who meet inclusion and exclusion criteria will be treated with EMB-001 (720 mg metyrapone/24 mg oxazepam mg BID, for a total daily dose of 1440 mg metyrapone and 48 mg oxazepam) for a 12-week period, followed by a one week taper.

During the Taper Period, subjects will receive EMB-001 240/8 mg BID.

There will be a follow-up visit for safety assessments at Week 15.

ELIGIBILITY:
Inclusion Criteria:

* Has signed the ICF and is able to read and understand the information provided in the ICF.
* Healthy smokers 21 to 65 years of age (inclusive) at screening.
* Smokes an average of at least 10 commercially available cigarettes per day for the last 12 months.
* Has an expired air CO reading of at least 10 ppm at screening.
* Express a desire to quit smoking within the next 30 days at screening.
* Serum Cortisol > 3 µg/dL at screening.
* Willing and able to comply with the requirements of the study.
* Owns a smart phone with text message and data capabilities compatible with necessary surveys.

Exclusion Criteria:

* Is unhealthy or cannot participate in the study for any reason (e.g., medical, psychiatric, and/or social reason) as judged by the Investigator or designated medical staff based on all available assessments from the screening period (e.g., safety laboratory, vital signs, physical examination, ECG, concomitant medications and medical history).
* PHQ-9 score greater than 9, or a score greater than 0 on item #9 ("Thoughts that you would be better off dead, or of hurting yourself in some way") at screening.
* Elevated aspartate aminotransferase (AST) or alanine aminotransferase (ALT) greater than two times the upper limit of normal or history of liver disease.
* Have positive serology test results for human immunodeficiency virus (HIV)-1/HIV-2 antibodies, hepatitis B surface antigen, or hepatitis C antibody.
* High blood pressure (systolic > 150 mmHg or diastolic >95 mmHg) at screening.
* Body mass index (BMI) less than 18.5 kg/m2 or greater than 35.0 kg/m2.
* Coronary heart disease, structural cardiac disease, cardiac dysrhythmias, abnormal ECG, syncope, cardiac chest pain, or history of heart attack or heart failure. For males, QTc > 450 msec. For females QTc > 470 msec (using Fridericia correction formula).
* Has a history of clinically significant drug/alcohol overdose as judged by the Investigator.
* Has alcohol breathalyzer > 0% at screening.
* Has a current DSM-5 opioid or benzodiazepine use disorder of any severity or use of these substances or alcohol in amounts that would increase risk of receiving oxazepam as part of EMB-001 or has received psychotherapy or behavioral treatments potentially impacting symptoms of depression, anxiety, or nicotine withdrawal within 30 days of screening, or during the study.
* Has history of mental illness that, in the opinion of the investigator, may interfere with subject safety or data integrity.
* Taking antidepressants, CNS or psychoactive medications (e.g., antipsychotics, benzodiazepines, hypnotics) or medications that prolong QTc within the last 30 days of screen or during study.
* Use of any of these products in the past 30 days:

  1. Illegal drugs (or if the urine drug screen is positive for cocaine, THC, amphetamines, methamphetamines, MDMA (Ecstasy), phencyclidine, benzodiazepines, barbiturates, or opiates at screening);
  2. Experimental (investigational) drugs or biologic;
  3. Chronic opiate use;
  4. Biotin products (Vitamin B7 or B8, Vitamin H, or coenzyme R).
* Use of glucocorticoids including:

  1. Oral glucocorticoids within 90 days of screen or during study;
  2. Inhaled glucocorticoids within 90 days of screen or during study;
  3. Topical glucocorticoids within 7 days of screen or during the study (except when applied to a small body surface area);
  4. Joint injection within 90 days of screening or during the study.
* Donation of any blood components within 84 days of screening or during the study or loss of blood ≥ 400 mL within 84 days of screen.
* Use of smokeless tobacco (chewing tobacco, snuff), cigars (except for cigarillos), pipes, hookah, e-cigarettes, nicotine replacement therapy or other smoking cessation treatments within 14 days of enrollment.
* Pregnant or nursing (by self-report) or has a positive pregnancy test.
* Woman of Childbearing Potential
* Known hypersensitivity to or intolerance of oxazepam, metyrapone, or any benzodiazepine, or severe hypersensitivity reaction (e.g., angioedema) to any drug.
* Treatment with an investigational drug or biologic within the 30 days preceding the first dose of study medication or plans to take another investigational drug or biologic within 30 days of study completion (including the follow-up visit).

Ages: 21 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2021-06-10 (Actual); Primary Completion 2023-04-01 (Actual); Study Completion 2023-05-01 (Actual)

PRIMARY OUTCOMES:
Smoking Abstinence | Weeks 9-12
  The primary abstinence outcome will be smoking abstinence

CONTACTS AND LOCATIONS:
Overall Officials: Bruce McCarthy, MD, Study Chair — Embera NeuroTherapeutics, Inc.
Locations (2):
- United States (2):
  - Embera Site, Miami Lakes, Florida
  - Rose Research Center, Raleigh, North Carolina

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Kablinger AS, Lindner MA, Casso S, Hefti F, DeMuth G, Fox BS, McNair LA, McCarthy BG, Goeders NE. Effects of the combination of metyrapone and oxazepam on cocaine craving and cocaine taking: a double-blind, randomized, placebo-controlled pilot study. J Psychopharmacol. 2012 Jul;26(7):973-81. doi: 10.1177/0269881111430745. Epub 2012 Jan 11. PMID 22236504